CLINICAL TRIAL: NCT01181856
Title: Safety and Immunogenicity of Candidate Tuberculosis (TB) Vaccine MVA85A Administered by the Intramuscular Route and the Intradermal Route: a Phase I Randomised Active Controlled Trial
Brief Title: Safety of Tuberculosis Vaccine, MVA85A, Administered by the Intramuscular Route and the Intradermal Route
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB022
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Tuberculosis
Keywords: Vaccine; MVA 85A
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Intramuscular immunisation
  Interventions: Biological: MVA 85A
- Group B (Experimental): Intradermal immunisation
  Interventions: Biological: MVA 85A

INTERVENTIONS:
Biological: MVA 85A — Single injection of 1 x 108 pfu MVA85A

SUMMARY:
This is a phase I study that will compare the safety and immunogenicity of candidate tuberculosis (TB) vaccine MVA85A administered by the intramuscular route and the intradermal route in healthy adult individuals who have been previously vaccinated with Bacillus Calmette-Guerin (BCG).

DETAILED DESCRIPTION:
We postulate that the intramuscular route is not inferior to the intradermal route of administration of MVA85A in BCG vaccinated adults when evaluated for safety and immunogenicity.

If MVA85A can be given safely by intramuscular route and it is at least equally immunogenic and efficacious in a prime-boost strategy, then it would probably be the preferred route in subsequent phase II and III trials. There are several reasons for this:

* Reduced pain associated with injection.
* Reduced local reaction at the injection site.
* More straightforward procedure; less technically demanding; less time consuming.
* Easier production and storage of vaccine.
* Larger volume of vaccine can be given.

Trials of MVA85A to date have established 1 x 10^8 pfu as the optimal dose for intradermal injection in adults. We therefore intend to administer this same dose intramuscularly in order to directly compare the two routes for both safety and immunogenicity. These results will guide future trials in which the intramuscular route, if safe, could be further evaluated at either higher or lower dose depending on immunogenicity at 1 x 10^8 pfu dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged 18 - 55 years (both male and female)
2. Resident in or near Oxford for the duration of the study period
3. Confirmation of prior vaccination with BCG not less than 3 months prior to projected study vaccination date (by visible BCG scar on examination or written documentation)
4. Normal medical history and physical examination
5. Willingness to allow the Investigators to discuss the individual's medical history with their GP
6. Willingness to use continuous effective barrier contraception for three months after receiving the vaccination (males and females)
7. Willingness to use effective contraception for the duration of the study period (females only)
8. Agreement to refrain from blood donation during the course of the study
9. Give written informed consent
10. Agreement to allow the Investigator to register volunteer details with a confidential database to prevent concurrent entry into clinical trials
11. Able and willing (in the Investigator's opinion) to comply with all the study requirements

Exclusion Criteria:

1. Clinical, radiological, or laboratory evidence of current active TB infection
2. Laboratory evidence at screening of latent TB infection as indicated by a positive ELISPOT test (greater than 17 sfc/million PBMC) in any ESAT6 peptide or CFP10 peptide poola
3. Previous vaccination with candidate vaccine MVA85A or another recombinant MVA vaccine
4. Clinically significant history of skin disorder, allergy, immunodeficiency (including human immunodeficiency virus [HIV]), cancer (except basal cell carcinoma [BCC] or carcinoma in situ [CIS]), cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
5. History of serious psychiatric condition
6. Concurrent oral or systemic steroid medication or the use of other immunosuppressive agents
7. History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the study vaccine
8. Any clinically significant abnormality of screening blood or urine tests
9. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) or HIV antibodies
10. Female currently lactating, confirmed pregnancy or intention to become pregnant during study period
11. Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device other than the study vaccine for 30 days prior to dosing with the study vaccine, or planned use during the study period
12. Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
13. Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the volunteer at risk or may influence the result of the study or may affect the volunteer's ability to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months following vaccination
  Safety data in both groups, as assessed by the frequency, incidence, and nature of adverse events (AEs) and serious adverse events (SAEs) during the study. Safety is measured throughout the 6 months follow up period, but specifically on the following days: 2, 7, 14, 28, 56, 84 and 168 and. Blood for safety testing is taken at Days 7 and 28.

SECONDARY OUTCOMES:
Immunogenicity | 6 months following vaccination
  Immunogenicity data in both groups. This will be obtained from exploratory immunological laboratory investigations on blood samples taken at screening, and throughout follow up. Immunogenicity is measured throughout the 6 months follow up period, but specifically on the following days: 2, 7, 14, 28, 56, 84 and 168.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- Centre of Clinical Vaccinology and Tropical Medicine (CCVTM) Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Meyer J, Harris SA, Satti I, Poulton ID, Poyntz HC, Tanner R, Rowland R, Griffiths KL, Fletcher HA, McShane H. Comparing the safety and immunogenicity of a candidate TB vaccine MVA85A administered by intramuscular and intradermal delivery. Vaccine. 2013 Feb 4;31(7):1026-33. doi: 10.1016/j.vaccine.2012.12.042. Epub 2012 Dec 21. PMID 23266342